CLINICAL TRIAL: NCT03880994
Title: Mental Health of Men Before and After Testicular Cancer Treatment. Danish: "Mænds Mentale Sundhed før og Efter Behandling af testikulær kræft"
Brief Title: Mental Health of Men Before and After Testicular Cancer Treatment
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: TC_Horsens
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-06

CONDITIONS: Testis Cancer; Cognitive Impairment; Sexual Dysfunction
Keywords: Sexual Health; Fatigue; Quality of Life; Depression; Anxiety; Fertility concerns; Sleep Quality; Erectile Function; Cognitive Impairment; Testis Cancer
MeSH Terms: conditions — Testicular Neoplasms; Cognitive Dysfunction; Sexual Dysfunction, Physiological; Fatigue; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study, that investigates men diagnosed with testicular cancer before and after treatment.

The patients are included at their visit at the Fertility clinic in Horsens, where they deposit semen for cryopreservation prior to surgery and potential systemic treatment. Here the patients, who want to participate will perform a cognitive test and afterwards complete a questioner (T1). After 9 month the patients will be invited to perform the cognitive test and complete the questionnaire again (T2).

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 - 45 years.
* Newly diagnosed testicular cancer and referred to the fertility clinic in Horsens fore cryopreservation of semen prior to further treatment.

Exclusion Criteria:

* Men, who cannot talk, read ore write Danish.
* Men who are not able to give informed consent.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men aged 18 - 45 years, with newly diagnosed testicular cancer referred to the fertility clinic in Horsens, Denmark, fore cryopreservation of semen prior to further treatment.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance, CANTAB iPad based cognitive performance test. | 9 months. The patients complete the cognitive test at baseline (T1) and again after 9 months (T2).
  The cognitive test is performed on an iPad using the validated Cambridge Neuropsychological Test Automated Battery (CANTAB) Connect Research software. The cognitive domains assessed are sensorimotor function and comprehension, processing and psychomotor speed, sustained attention, visual episodic memory, working memory and strategy, visual working memory and planning, each at T1 and T2. Comparison of test results from T1 and T2 will assess if there is a change in the cognitive performance.
Change in Self reported Cognitive Performance | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  Assessed by The Patients Assessment of Own Functioning Inventory (PAOFI)
Change in Sexual Health | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  Assessed by the EORTC Sexual Health Questionnaire (EORTC SHQ-C22)
Change in Erectile Function | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  Assessed by The International Index of Erectile Function (IIEF-5)
Change in symptoms of Depression and Anxiety | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  Assessed by the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item scale with 2 subscales measuring severity of anxiety (HADS-A) and depression (HADS-D) symptoms. Each subscale has 7 items and each item is scored from 0-3. Thus, the total score for each subscale range from 0-21, with 0 indicating no symptoms and 21 severe symptoms.
Change in Fatigue | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  Assessed by the FACIT_Fatigue Questionnaire. The questionnaire consists of 13-items each scored from 0-4. The scores are summarized, and the total score range from 0-52 with higher score denoting less fatigue.
Change in Sleep Quality | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  Assessed by the Pittsburgh Sleep Quality Index (PSQI)

SECONDARY OUTCOMES:
Change in Quality of Life | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  The quality of life is assessed by a subscale from the WHO Quality of Life (WHOQOL)-BREF questionnaire. The subscale has 2 questions each scored from 1-5. Thus, the total score for this subscale range from 2-10 with higher scores denoting higher quality of life.
Change in Well being | 9 months. The patients complete the questionnaire at baseline (T1) and again after 9 months (T2).
  The wellbeing is assessed by the WHO (Five) Well-being scale (WHO-5), that has 5 questions each scored from 0-5. The raw score ranges from 0-25 and is multiplied by 4 to give the final score that ranges from 0-100, with higher scores denoting higher wellbeing.
Fertility related concerns | The Patients complete the questions at baseline (T1).
  The patient answers 5 questions regarding fertility related concerns, investigating if he has concerns about being able to become a father with or without fertility assistance. Also, the patient answers 4 questions regarding the information given by healthcare professionals, to assess if he finds, that he has been given enough information regarding semen deposit and possible later fertility assistance.
  None of these 9 questions are validated.

CONTACTS AND LOCATIONS:
Locations (1):
- Horsens fertility Clinic, Region Hospital Horsens, Horsens, Denmark

REFERENCES:
- [Derived] Hojris NF, Frederiksen Y, Agerbaek M, Nielsen SH, Holt M, Brand SL, Petersen NL, Knudsen UB, Amidi A. Longitudinal assessment of cognitive function in testicular cancer patients prior to orchiectomy and 9 months later and associations with tumor markers. Support Care Cancer. 2025 Jun 17;33(7):591. doi: 10.1007/s00520-025-09637-w. PMID 40526183